CLINICAL TRIAL: NCT01961076
Title: New Approaches for Over-night Feeding in Glycogen Storage Disease Type 1 (GSD 1)
Brief Title: Overnight Feeding Study in Glycogen Storage Disease Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2013-0161
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Glycogen Storage Disease Type 1 (GSD 1)
MeSH Terms: conditions — Glycogen Storage Disease Type I

ARMS (3):
- uncooked corn starch (Experimental): Patients receive uncooked corn starch before bed-time
  Interventions: Other: overnight nutrition regime
- modified corn starch (Experimental): Patients receive modified corn starch before bed-time
  Interventions: Other: overnight nutrition regime
- other carbohydrate (starch) containing meal (Experimental): Patients receive a carbohydrate (starch) containing meal before bed-time
  Interventions: Other: overnight nutrition regime

INTERVENTIONS:
Other: overnight nutrition regime — Patients receive the specified overnight nutrition regimen

SUMMARY:
In this clinical cross-over study, we will compare the efficacy of different oral nutrition regimens for night-time glucose control in adult GSD 1 patients. Three different over-night nutrition regimens (=interventions) will be compared in each patient sequentially, (1) uncooked corn starch (UCSS, "Maizena"), (2) modified corn-starch, (3) other carbohydrate (starch) containing meal. During each intervention, glucose profiles will be continuously monitored by continuous glucose monitoring (CGMS). The duration of each intervention is 3d (mimimum) to 6d (maximum), depending on the quality of night-time glucose control and the technical quality of glucose sensor readings. Between the interventions, the patients follow their normal prescribed diet.

ELIGIBILITY:
Inclusion criteria:

* Glycogen storage disease type 1 (type 1a and 1b)
* Stable nighttime glucose control without frequent or severe hypoglycaemia under current dietary treatment, according to capillary glucose measurements.

Exclusion criteria:

* Unstable night-time glucose control during the last 8 weeks with frequent (> 4x weekly) hypoglycaemia during night-time, or a hospitalisation due to unstable glucose control during the last 4 weeks, or any episode of severe hypoglycaemia (requiring assistance or loss of consciousness) during the last 4 weeks.
* Pregnancy or breast feeding
* Drug or alcohol abuse
* Acute gastrointestinal problems (e.g. acute gastroenteritis)
* Known malignancy (e.g. hepatocellular carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum fasting time over-night (h) | Maximum fasting time will be measured during each dietary intervention for an average period of 3d (minimum) to 6d (maximum)

CONTACTS AND LOCATIONS:
Overall Officials: Giatgen Spinas, Prof MD, Principal Investigator — University Hospital Zurich, Division of Endocrinology, Diabetes and Clinical Nutrition
Locations (1):
- University Hospital Zurich, Division of Endocrinology, Diabetes and Clinical Nutrition, Zurich, Canton of Zurich, Switzerland